CLINICAL TRIAL: NCT03441360
Title: A Phase 2, Multicenter, Open-label Study to Assess Safety and Preliminary Activity of Eribulin Mesylate in Pediatric Subjects With Relapsed/Refractory Rhabdomyosarcoma (RMS), Non-rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS) and Ewing Sarcoma (EWS)
Brief Title: Study to Assess Safety and Preliminary Activity of Eribulin Mesylate in Pediatric Participants With Relapsed/Refractory Rhabdomyosarcoma (RMS), Non-rhabdomyosarcoma Soft Tissue Sarcoma (NRSTS) and Ewing Sarcoma (EWS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7389-G000-223
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Results first posted 2022-01-28 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-01

CONDITIONS: Relapsed/Refractory Rhabdomyosarcoma; Non-rhabdomyosarcoma Soft Tissue Sarcoma; Ewing Sarcoma
Keywords: eribulin mesylate; pediatric
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma; Sarcoma, Ewing | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Eribulin mesylate 1.4 mg/m^2: RMS (Experimental): Pediatric participants with relapsed/refractory rhabdomyosarcoma (RMS) will receive eribulin mesylate administered as an intravenous (IV) infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 milligrams per meters squared (mg/m^2). Participants will continue study therapy until progression of disease (per Response Evaluation Criteria In Solid Tumors [RECIST] 1.1), intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Eribulin mesylate
- Eribulin mesylate 1.4 mg/m^2: NRSTS (Experimental): Pediatric participants with non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) will receive eribulin mesylate administered as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants will continue study therapy until progression of disease (per RECIST 1.1), intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Eribulin mesylate
- Eribulin mesylate 1.4 mg/m^2: EWS (Experimental): Pediatric participants with Ewing sarcoma (EWS) will receive eribulin mesylate administered as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants will continue study therapy until progression of disease (per RECIST 1.1), intolerable toxicity, or withdrawal of consent.
  Interventions: Drug: Eribulin mesylate

INTERVENTIONS:
Drug: Eribulin mesylate — Intravenous infusion

SUMMARY:
This study will be conducted as an assessment of the safety and preliminary activity of eribulin mesylate in pediatric participants with relapsed/refractory rhabdomyosarcoma (RMS), non-rhabdomyosarcoma soft tissue sarcoma (NRSTS), or Ewing sarcoma (EWS) to determine whether each cohort warrants further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥12 months to <18 years old at the time of informed consent
* Diagnosis: Histologically confirmed rhabdomyosarcoma (RMS), non-rhabdomyosarcoma soft tissue sarcoma (NRSTS) (Grade 2 or 3), or Ewing sarcoma (EWS) which is relapsed or refractory (failed front line therapy)
* The presence of measurable disease meeting the following criteria:

  * At least 1 lesion of ≥1.0 centimeter (cm) in the longest diameter for a non-lymph node or ≥1.5 cm in the short-axis diameter for a lymph node that is serially measurable according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 using computerized tomography/magnetic resonance imaging (CT/MRI).
  * Lesions that have had radiotherapy must show subsequent radiographic evidence of increase in size by at least 20% to be deemed a target lesion.
* Therapeutic options: Participant's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life.
* Performance level: Performance score ≥50%. Karnofsky (for participants >16 years of age) or Lansky (for participants ≤16 years of age). Participants who are unable to walk because of paralysis and/or previous surgeries, but who are in a wheelchair, will be considered ambulatory for the purpose of assessing performance score.
* Participants must have fully recovered from the acute toxic effects of all prior anticancer therapy and must meet the following minimum duration from prior anticancer directed therapy prior to study drug administration. If, after the required time frame, the numerical eligibility criteria are met, eg, blood count criteria, the participant is considered to have recovered adequately:

  * Cytotoxic chemotherapy or other chemotherapy known to be myelosuppressive: ≥21 days after the last dose of cytotoxic or myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * Anticancer agents not known to be myelosuppressive (eg, not associated with reduced platelet or absolute neutrophil count [ANC] counts): ≥7 days after the last dose of agent.
  * Monoclonal antibodies ≥ 3 half-lives must have elapsed from infusion of last dose of antibody (including checkpoint inhibitors), and toxicity related to prior antibody therapy must be recovered to Grade ≤1.
  * Hematopoietic growth factors: ≥14 days after the last dose of a long-acting growth factor (eg, Neulasta) or 7 days for a short-acting growth factor. For agents that have known adverse events (AEs) occurring beyond 7 days after administration, this period must be extended beyond the time during which AEs are known to occur. The duration of this interval must be discussed with the sponsor.
  * Interleukins, interferons, and cytokines (other than hematopoietic growth factors): ≥21 days after the completion of interleukins, interferons, or cytokines (other than hematopoietic growth factors)
  * Stem cell infusions (with or without total body irradiation [TBI]): ≥84 days
  * Allogeneic (non-autologous) bone marrow or stem cell transplant, or any stem cell infusion including donor lymphocyte infusion or boost infusion: ≥84 days after infusion and no evidence of graft versus host disease (GVHD)
  * Autologous stem cell infusion including boost infusion: ≥42 days
  * Cellular therapy: ≥42 days after the completion of any type of cellular therapy (eg, modified T-cells, natural killer cells, dendritic cells, etc)
  * Radiation therapy (XRT)/External Beam Irradiation including Protons: ≥14 days after local XRT; ≥150 days after TBI, craniospinal XRT or if radiation to ≥50% of the pelvis; ≥42 days if other substantial BM radiation
  * Radiopharmaceutical therapy (eg, radiolabeled antibody, 131I-metaiodobenzylguanidine): ≥42 days after systemically administered radiopharmaceutical therapy.
* Adequate bone marrow function, defined as:

  * ANC ≥1.0 × 10^9/Liter (L)
  * Platelet count ≥100 × 10^9/L (transfusion independent, defined as not receiving platelet transfusions within a 7-day period prior to study drug administration)
  * Hemoglobin at least 8.0 grams per deciliter (g/dL) at Baseline (blood transfusions are allowed during the screening period to correct hemoglobin values less than 8.0 g/dL) Note: As blood transfusions are permitted to meet the hemoglobin criteria, participants requiring transfusion must not be known to be refractory to red blood cell or platelet transfusions.
* Adequate renal function, defined as:

  * A serum creatinine based on age/gender, derived from the Schwartz formula for estimating glomerular filtration rate (GFR)
  * Or creatinine clearance or GFR ≥50 milliliters per minute (mL/min)/1.73 meters squared (m^2) based on a 12 or 24 hour urine creatinine collection
* Adequate liver function, defined as:

  * Bilirubin (sum of conjugated + unconjugated) ≤1.5 × upper limit of normal (ULN) for age
  * Alanine aminotransferase (ALT) ≤110 units per Liter (U/L). For the purpose of this study, the ULN for ALT is 45 U/L
  * Serum albumin ≥2 g/dL
* Informed consent: All participants and/or their parents or legally authorized representatives must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines. Participants must be willing to comply with all aspects of the protocol.

Exclusion Criteria:

* Pregnancy, breastfeeding, contraception: Females who are breastfeeding or pregnant at Screening or Baseline (as documented by a positive beta-human chorionic [β-hCG] or human chorionic gonadotropin [hCG] test with a minimum sensitivity of 25 International Units per Liter [IU/L] or equivalent units of β-hCG [or hCG]). A separate baseline assessment is required if a negative screening pregnancy test was obtained more than 72 hours before the first dose of study drug.

  * Females of childbearing potential (all post pubertal females will be considered to be of childbearing potential unless they have early menopause [amenorrheic for at least 12 consecutive months, in the appropriate age group, and without other known or suspected cause] or have been sterilized surgically [ie, bilateral tubal ligation, total hysterectomy, or bilateral oophorectomy, all with surgery at least 1 month before dosing]) who:
  * Do not agree to use a highly effective method of contraception for the entire study period and for 6 months after study drug discontinuation, ie:
  * Total abstinence (if it is their preferred and usual lifestyle);
  * An intrauterine device (IUD) or intrauterine system (IUS);
  * A contraceptive implant;
  * An oral contraceptive (must be on a stable dose of the same oral hormonal contraceptive product for at least 4 weeks before dosing with study drug and for the duration of the study and for 6 months after study drug discontinuation); or
  * Do not have a vasectomized partner with confirmed azoospermia.

For sites outside of the European Union (EU), it is permissible that if a highly effective method of contraception is not appropriate or acceptable to the participant, or the participant has commenced/adjusted/changed oral hormonal contraceptive product/dose within 4 weeks prior to study drug administration, then the participant must agree to use a medically acceptable method of contraception, ie, double barrier methods of contraception such as condoms plus diaphragm or cervical/vault cap with spermicide.

* Males who have not had a successful vasectomy (confirmed azoospermia) or if they and their female partners do not meet the criteria above (ie, not of childbearing potential or practicing highly effective contraception throughout the study period or for 3 months after study drug discontinuation). No sperm donation is allowed during the study period or for 3 months after study drug discontinuation.

  - Concomitant medications:
* Corticosteroids: Participants receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to study drug administration (except when indicated for Central Nervous System [CNS] metastases, then participants must not have received corticosteroids for at least 28 days)
* Anticancer Agents: participants who are currently receiving other anticancer agents
* Anti-GVHD agents Post-transplant: Participants who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant
* Strong CYP3A4 inducers/inhibitors

  * Received prior therapy with eribulin mesylate
  * Any other malignancy that required treatment (except for non-melanoma skin cancer, or histologically confirmed complete excision of carcinoma in situ), within 2 years prior to study drug administration
  * Has hypersensitivity to eribulin or any of the excipients
  * Has a prior history of viral hepatitis (B or C) as demonstrated by positive serology (presence of antigens) or have an uncontrolled infection requiring treatment. Participants with a known prior history of hepatitis B or C may be eligible pending agreement with the sponsor.
  * Has > Grade 1 peripheral sensory neuropathy or > Grade 1 peripheral motor neuropathy graded according to the Modified ("Balis") Pediatric Scale of Peripheral Neuropathies
  * Has cardiac pathology: Participants with known congestive heart failure, symptomatic or left ventricular (LV) ejection fraction <50% or shortening fraction <27%
  * Participants with congenital long QT syndrome, bradyarrhythmias, or QTc >480 millisecond (msec) on at least 2 separate electrocardiograms (ECGs).
  * Has CNS Disease: Participants with brain or subdural metastases are not eligible unless the metastases are asymptomatic and do not require treatment or have been adequately treated by local therapy (eg, surgery or radiotherapy) and have discontinued the use of corticosteroids for this indication for at least 4 weeks prior to study drug administration. Confirmation of radiographic stability must be done by comparing the brain scan (CT or MRI) performed during the Screening Period, using the same imaging modality, to a brain scan performed earlier (and following local therapy where applicable). Participants must be clinically stable. It is not the intention of this protocol to treat participants with active brain metastases.

Note: CNS imaging is required to confirm eligibility for participants with a known history of CNS disease.

* Have had or are planning to have the following invasive procedures:

  * Major surgical procedure or significant traumatic injury within 28 days prior to study drug administration
  * Laparoscopic procedure or open biopsy within 7 days prior to study drug administration
  * Central line placement or subcutaneous port placement is not considered major surgery but must be placed at least 2 days prior to study drug administration
  * Core biopsy, including bone marrow biopsy, within 2 days prior to study drug administration
  * Fine needle aspirate within 3 days prior to study drug administration
* Has any serious concomitant illness that in the opinion of the investigator(s) could affect the participant's safety or interfere with the study assessments
* Participants with known human immunodeficiency virus (HIV); due to lack of available safety data for eribulin therapy in HIV-infected participants

Ages: 12 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2022-01-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Loma Linda University Cancer Center, Loma Linda, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Southern California Permanente Medical Group, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital- San Diego, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Nemours / A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nemours Children's Clinic, Jacksonville, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children - Indiana University, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Norton Children's Hospital, Louisville, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - CS Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospital and Clinics, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Rutgers cancer Institute of NJ, New Brunswick, New Jersey
  - Columbia University Medical Center, New York, New York
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Randall Children's Hospital at Legacy Emanuel, Portland, Oregon
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Health Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - Children's Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Children's Hosptial of The King's Daughters, Norfolk, Virginia
  - Seattle Children's, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 38 investigative sites in the United States from 17 April 2018 to 21 January 2022.
Pre-assignment Details: A total of 24 participants were screened, of which 1 was screen failure and 23 participants were enrolled, out of which 21 participants were randomized and treated in the study and 2 were not treated due to withdrawal of consent and rapid disease progression (1 participant from each arm).
Groups:
- Eribulin Mesylate 1.4 mg/m^2: RMS: Pediatric participants with rhabdomyosarcoma (RMS) received eribulin mesylate as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 milligrams per meter square (mg/m^2). Participants continued to receive study therapy until progression of disease, per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1), exhibited no clinical benefit, intolerable toxicity, withdrawal of consent or termination of the study program, whichever occurred first.
- Eribulin Mesylate 1.4 mg/m^2: NRSTS: Pediatric participants with non-rhabdomyosarcoma solid tumor sarcoma (NRSTS) received eribulin mesylate as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants continued to receive study therapy until progression of disease, (per RECIST 1.1), exhibited no clinical benefit, intolerable toxicity, withdrawal of consent or termination of the study program, whichever occurred first.
- Eribulin Mesylate 1.4 mg/m^2: EWS: Pediatric participants with Ewing sarcoma (EWS) received eribulin mesylate as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants continued to receive study therapy until progression of disease, (per RECIST 1.1), exhibited no clinical benefit, intolerable toxicity, withdrawal of consent or termination of the study program, whichever occurred first.
Period: Overall Study
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Started | 8 | 8 | 5
Completed | 0 | 0 | 0
Not Completed | 8 | 8 | 5
Not completed — Radiological disease progression | 5 | 6 | 4
Not completed — Clinical disease progression | 2 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who receive at least 1 dose of study drug.
Groups:
- Eribulin Mesylate 1.4 mg/m^2: RMS: Pediatric participants with RMS received eribulin mesylate as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants continued to receive study therapy until progression of disease, (per RECIST 1.1), exhibited no clinical benefit, intolerable toxicity, withdrawal of consent or termination of the study program, whichever occurred first.
- Eribulin Mesylate 1.4 mg/m^2: EWS: Pediatric participants with EWS received eribulin mesylate as an IV infusion on Days 1 and 8 of each 21-day cycle at a dose of 1.4 mg/m^2. Participants continued to receive study therapy until progression of disease, (per RECIST 1.1), exhibited no clinical benefit, intolerable toxicity, withdrawal of consent or termination of the study program, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS | Total
Number analyzed (Participants) | 8 | 8 | 5 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.4 (4.53) | 11.8 (5.57) | 13.2 (4.32) | 11.6 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 1 | 7
  Male | 6 | 4 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 6
  Not Hispanic or Latino | 5 | 6 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 5
  White | 5 | 4 | 2 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants achieving a best objective response of partial response (PR) or complete response (CR) per RECIST 1.1, by up to 24 weeks after all participants have completed response assessment. Response assessment was determined by investigator. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to less than (<) 10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From date of randomization up to first documentation of disease progression (PD) or date of death, whichever occurred first (approximately 32 months)
Population: The FAS included all participants who receive at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
percentage of participants | 0 [0.0 to 36.9] | 0 [0.0 to 36.9] | 0 [0.0 to 52.2]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the first dose date to the date of PD or date of death (whichever occurred first). PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions was also considered progression). Data for this secondary endpoint was collected and analyzed up to the primary completion date (PCD). As there was no further data collected, therefore data is reported till PCD only.
Time Frame: From the time from the first dose date to the date of disease progression (PD) or date of death, whichever occurred first (up to approximately 32 months)
Population: The FAS included all participants who receive at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
months | 1.74 [1.12 to 2.86] | 1.30 [0.62 to 1.51] | 0.76 [0.59 to 4.04]

3. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in participant administered with an investigational product. An SAE was any untoward medical occurrence that at any dose: resulted in death; life threatening; requires participant hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; was a congenital anomaly/birth defect (in the child of a participant who was exposed to the study drug). A treatment-emergent adverse event (TEAE) was defined as an AE that emerges during treatment, having been absent at pretreatment (Baseline) or (1) reemerges during treatment, having been present at pretreatment (Baseline) but stopped before treatment, or (2) worsens in severity during treatment relative to the pretreatment state, when the AE is continuous.
Time Frame: From date of administration of first dose up to 28 days after the last dose, or until resolution, whichever came first (up to approximately 45 months)
Population: The safety analysis set included all participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
Participants
  TEAEs | 8 | 8 | 5
  SAEs | 6 | 2 | 3

4. Secondary Outcome: Number of Participants With a Shift From Baseline to Worst Post-Baseline Common Terminology Criteria for Adverse Events (CTCAE) Grade in Laboratory Value
Description: Laboratory results were graded using CTCAE Version 4.03. As per CTCAE, Grade 1 scales as Mild; Grade 2 scales as Moderate; Grade 3 scales as severe or medically significant but not immediately life threatening; Grade 4 scales as life-threatening consequences. Data for this secondary endpoint was collected and analyzed up to the PCD. As there was no further data collected, therefore data is reported till PCD only.
Time Frame: From first dose of study drug up to approximately 32 months
Population: The safety analysis set included all participants who receive at least 1 dose of study drug. Here number analyzed "n" are the participants who were evaluable for the outcome measure for given categories with non-missing data at both baseline and any post-baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
Participants
  Baseline to Worst Post-baseline Grade 0, Hemoglobin Decreased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 1, Hemoglobin Decreased | 3 | 4 | 3
  Baseline to Worst Post-baseline Grade 2, Hemoglobin Decreased | 0 | 1 | 2
  Baseline to Worst Post-baseline Grade 3, Hemoglobin Decreased | 5 | 3 | 0
  Baseline to Worst Post-baseline Grade 4, Hemoglobin Decreased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 0, Hemoglobin increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 1, Hemoglobin increased | 0 | 0 | 0
  Worst Post-Baseline Grade 2, Hemoglobin increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 3, Hemoglobin increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 4, Hemoglobin increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 0, White blood cells decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 0, White blood cells decreased | 0 | 1 | 0
  Baseline to Worst Post-baseline Grade 1, White blood cells decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 1, White blood cells decreased | 4 | 2 | 1
  Baseline to Worst Post-baseline Grade 2, White blood cells decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 2, White blood cells decreased | 2 | 1 | 0
  Baseline to Worst Post-baseline Grade 3, White blood cells decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 3, White blood cells decreased | 0 | 2 | 3
  Baseline to Worst Post-baseline Grade 4, White blood cells decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 4, White blood cells decreased | 2 | 1 | 1
  Baseline to Worst Post-baseline Grade 0, White blood cells increased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 0, White blood cells increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 1, White blood cells increased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 1, White blood cells increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 2, White blood cells increased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 2, White blood cells increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 3, White blood cells increased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 3, White blood cells increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 4, White blood cells increased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 4, White blood cells increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 0, Lymphocyte count decreased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 0, Lymphocyte count decreased | 3 | 2 | 0
  Baseline to Worst Post-baseline Grade 1, Lymphocyte count decreased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 1, Lymphocyte count decreased | 1 | 0 | 0
  Baseline to Worst Post-baseline Grade 2, Lymphocyte count decreased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 2, Lymphocyte count decreased | 1 | 0 | 3
  Baseline to Worst Post-baseline Grade 3, Lymphocyte count decreased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 3, Lymphocyte count decreased | 2 | 4 | 2
  Baseline to Worst Post-baseline Grade 4, Lymphocyte count decreased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 4, Lymphocyte count decreased | 1 | 0 | 0
  Baseline to Worst Post-baseline Grade 0, Lymphocyte count increased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 0, Lymphocyte count increased | 8 | 4 | 5
  Baseline to Worst Post-baseline Grade 1, Lymphocyte count increased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 1, Lymphocyte count increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 2, Lymphocyte count increased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 2, Lymphocyte count increased | 0 | 2 | 0
  Baseline to Worst Post-baseline Grade 3, Lymphocyte count increased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 3, Lymphocyte count increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 4, Lymphocyte count increased: number analyzed (Participants) | 8 | 6 | 5
  Baseline to Worst Post-baseline Grade 4, Lymphocyte count increased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 0, Neutrophil count decreased: number analyzed (Participants) | 7 | 7 | 5
  Baseline to Worst Post-baseline Grade 0, Neutrophil count decreased | 1 | 0 | 1
  Baseline to Worst Post-baseline Grade 1, Neutrophil count decreased: number analyzed (Participants) | 7 | 7 | 5
  Baseline to Worst Post-baseline Grade 1, Neutrophil count decreased | 1 | 0 | 0
  Baseline to Worst Post-baseline Grade 2, Neutrophil count decreased: number analyzed (Participants) | 7 | 7 | 5
  Baseline to Worst Post-baseline Grade 2, Neutrophil count decreased | 3 | 1 | 0
  Baseline to Worst Post-baseline Grade 3, Neutrophil count decreased: number analyzed (Participants) | 7 | 7 | 5
  Baseline to Worst Post-baseline Grade 3, Neutrophil count decreased | 0 | 1 | 3
  Baseline to Worst Post-baseline Grade 4, Neutrophil count decreased: number analyzed (Participants) | 7 | 7 | 5
  Baseline to Worst Post-baseline Grade 4, Neutrophil count decreased | 2 | 5 | 1
  Baseline to Worst Post-baseline Grade 0, Platelet count decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 0, Platelet count decreased | 5 | 6 | 3
  Baseline to Worst Post-baseline Grade 1, Platelet count decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 1, Platelet count decreased | 2 | 1 | 2
  Baseline to Worst Post-baseline Grade 2, Platelet count decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 2, Platelet count decreased | 1 | 0 | 0
  Baseline to Worst Post-baseline Grade 3, Platelet count decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 3, Platelet count decreased | 0 | 0 | 0
  Baseline to Worst Post-baseline Grade 4, Platelet count decreased: number analyzed (Participants) | 8 | 7 | 5
  Baseline to Worst Post-baseline Grade 4, Platelet count decreased | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Electrocardiogram (ECG) Values
Description: Data for this secondary endpoint was collected and analyzed up to the PCD. As there was no further data collected, therefore data is reported till PCD only.
Time Frame: From first dose of study drug up to approximately 32 months
Population: The safety analysis set included all participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values
Description: as for outcome 5
Time Frame: From first dose of study drug up to approximately 32 months
Population: The safety analysis set included all participants who receive at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
Participants | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline for Lansky Play-performance Scale
Description: Reduced activities of daily living was assessed using the Lansky Play Performance Scale, where 100=fully active; 90=minor restrictions in strenuous physical activity; 80=active, gets tired more quickly; 70=greater restriction of play, less time spent in play activity; 60=up and around, active play minimal; quieter activities; 50=lying around much of the day; no active playing, all quiet play and activities; 40=mainly in bed; quiet activities; 30=bedbound; needs assistance even for quiet play; 20=sleeps often; play limited to very passive activities; 10=doesn't play or get out of bed; 5=unresponsive 0=dead. Data for this secondary endpoint was collected and analyzed up to the PCD. As there was no further data collected, therefore data is reported till PCD only.
Time Frame: Baseline up to approximately 32 months
Population: The safety analysis set included all participants who receive at least 1 dose of study drug. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure with non-missing data at both baseline and any post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 7 | 7 | 4
Participants
  Baseline score 70 to worst post-baseline score 50 | 1 | 0 | 0
  Baseline score 70 to worst post-baseline score 60 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 70 | 2 | 0 | 1
  Baseline score 70 to worst post-baseline score 80 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 90 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 100 | 0 | 0 | 0
  Baseline score 80 to worst post-baseline score 50 | 0 | 0 | 0
  Baseline score 80 to worst post-baseline score 60 | 1 | 0 | 0
  Baseline score 80 to worst post-baseline score 70 | 1 | 1 | 0
  Baseline score 80 to worst post-baseline score 80 | 0 | 2 | 1
  Baseline score 80 to worst post-baseline score 90 | 0 | 0 | 0
  Baseline score 80 to worst post-baseline score 100 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 50 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 60 | 0 | 0 | 1
  Baseline score 90 to worst post-baseline score 70 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 80 | 1 | 0 | 1
  Baseline score 90 to worst post-baseline score 90 | 0 | 2 | 0
  Baseline score 90 to worst post-baseline score 100 | 0 | 0 | 0
  Baseline score 100 to worst post-baseline score 50 | 0 | 0 | 0
  Baseline score 100 to worst post-baseline score 60 | 0 | 0 | 0
  Baseline score 100 to worst post-baseline score 70 | 1 | 1 | 0
  Baseline score 100 to worst post-baseline score 80 | 0 | 0 | 0
  Baseline score 100 to worst post-baseline score 90 | 0 | 0 | 0
  Baseline score 100 to worst post-baseline score 100 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Shift From Baseline to Worst Post-baseline for Karnofsky Performance Status Scores
Description: Karnofsky performance status assessed as best and worst score change from baseline using Karnofsky performance criteria.Score classified participants based on functional impairment. Ranges from 0-100, lower score, worst survival for most serious illnesses, 100=normal;no complaints;no evidence of disease;90=able to carry on normal activity with effort,minor sign or symptoms of disease;80=normal activity with effort;some sign or symptoms of disease;70= cares for self;unable to carry on normal activity or do active work;60=requires occasional assistance,but able to care for most personal needs;50=requires considerable assistance;frequent medical care;40=disabled;requires special care; assistance;30=severely disabled;hospitalization indicated,although death is not imminent;20=very sick;hospitalization; 10=moribund;fatal processes progressively worsening;0=dead.Data for this endpoint was collected;analyzed up to PCD. As no further data collected, therefore data is reported till PCD only.
Time Frame: Baseline up to approximately 32 months
Population: The safety analysis set included all participants who receive at least 1 dose of study drug. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure for the outcome measure with non-missing data at both baseline and any post-baseline timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 1 | 0 | 1
Participants
  Baseline score 70 to worst post-baseline score 50 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 60 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 70 | 1 | 0 | 0
  Baseline score 70 to worst post-baseline score 80 | 0 | 0 | 0
  Baseline score 70 to worst post-baseline score 90 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 50 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 60 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 70 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 80 | 0 | 0 | 1
  Baseline score 90 to worst post-baseline score 90 | 0 | 0 | 0
  Baseline score 90 to worst post-baseline score 100 | 0 | 0 | 0

9. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the time from the first date of documented PR or CR to the date of disease progression or date of death (whichever occurred first). CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must had reduction in the short axis to <10 mm. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study). Data for this secondary endpoint was collected and analyzed up to the PCD. As there was no further data collected, therefore data is reported till PCD only.
Time Frame: From day of first documentation of PR or CR to the day of disease progression or death (up to approximately 32 months)
Population: The FAS included all participants who receive at least 1 dose of study drug. Here overall number analyzed "N" are the participants who were evaluable for the outcome measure however no participant with complete response or partial response were observed in this study.
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the first dose date to the date of death.
Time Frame: From the day of first dose to the day of death, up to approximately 45 months
Population: The FAS included all participants who receive at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
Number analyzed (Participants) | 8 | 8 | 5
months | 5.08 [1.74 to 6.47] | 6.95 [0.72 to 16.26] | 7.89 [2.50 to 29.80]

ADVERSE EVENTS:
Time Frame: From date of administration of first dose up to 28 days after the last dose, or until resolution, whichever came first (up to approximately 45 months)
Arm/Group | Eribulin Mesylate 1.4 mg/m^2: RMS | Eribulin Mesylate 1.4 mg/m^2: NRSTS | Eribulin Mesylate 1.4 mg/m^2: EWS
All-Cause Mortality (participants affected / at risk) | 8/8 | 7/8 | 5/5
Serious Adverse Events (participants affected / at risk) | 6/8 | 2/8 | 3/5
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2: RMS (N=8) | Eribulin Mesylate 1.4 mg/m^2: NRSTS (N=8) | Eribulin Mesylate 1.4 mg/m^2: EWS (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eribulin Mesylate 1.4 mg/m^2: RMS (N=8) | Eribulin Mesylate 1.4 mg/m^2: NRSTS (N=8) | Eribulin Mesylate 1.4 mg/m^2: EWS (N=5)
Anaemia (Blood and lymphatic system disorders) | 5 (24) | 5 (7) | 4 (16)
Leukopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (6) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (3) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (3) | 2 (2) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7) | 1 (1) | 1 (1)
Face oedema (General disorders) | 1 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (8) | 4 (4) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 3 (3) | 2 (2)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 2 (3) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 5 (9) | 2 (2) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 6 (12) | 1 (3) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 2 (3) | 2 (3) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (4) | 1 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 1 (1) | 2 (3)
International normalised ratio increased (Investigations) | 1 (3) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (9) | 4 (5) | 3 (13)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 7 (13) | 4 (11) | 4 (26)
Platelet count decreased (Investigations) | 2 (4) | 1 (2) | 2 (3)
Protein urine present (Investigations) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 0 (0) | 0 (0)
Weight increased (Investigations) | 1 (4) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 6 (16) | 4 (12) | 3 (23)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (12) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 (10) | 1 (1) | 2 (4)
Hypocalcaemia (Metabolism and nutrition disorders) | 3 (6) | 0 (0) | 1 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 3 (3) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 3 (5) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (3) | 2 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (10) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tracheal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 4 (4) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 4 (5) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT03441360/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03441360/SAP_002.pdf